CLINICAL TRIAL: NCT07322848
Title: Drug Eluting Beads Transarterial Chemoembolization Versus Conventional Transarterial Chemoembolization for Beyond-Milan-Criteria Hepatocellular Carcinoma After Transjugular Intrahepatic Portosystemic Shunt: A Phase 3, Open Label, Multicenter, Randomized Controlled Trial
Brief Title: DEB-TACE vs cTACE in HCC After TIPS
Acronym: UPGRADE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jiaping Li, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2025]634
Record Dates: First submitted 2025-12-04; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma (HCC); TACE; TIPS; DEB-TACE; cTACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB-TACE group (Experimental)
  Interventions: Procedure: DEB-TACE
- cTACE group (Experimental)
  Interventions: Procedure: cTACE

INTERVENTIONS:
Procedure: DEB-TACE — Experienced interventional radiologists perform transarterial chemoembolization using drug-eluting microspheres (100-300 μm or 300-500 μm) loaded with chemotherapeutic agents (e.g., 70 mg epirubicin or doxorubicin). The procedure involves superselective catheterization of tumor-feeding arteries, with embolization endpoint being angiographic stasis of arterial flow. Repeat treatments are based on 6-8 week imaging, if residual active lesions and preserved liver function are present. Treatment is discontinued upon disease progression, non-operable conditions, or persistent liver impairment.
  Arms: DEB-TACE group
Procedure: cTACE — Patients receive conventional transarterial chemoembolization using ethiodized oil loaded with chemotherapeutic agents (e.g., 40 mg epirubicin or doxorubicin) followed by gelatin sponge particle embolization if needed. Procedures are performed by experienced interventional radiologists with superselective catheterization. Repeat treatments are based on 6-8 week imaging, provided liver function is preserved. Treatment stops upon disease progression, vascular inoperability, or sustained liver impairment.
  Arms: cTACE group

SUMMARY:
This is a Phase 3, open-label, multicenter, randomized controlled clinical trial designed to evaluate the efficacy and safety of Drug-Eluting Bead Transarterial Chemoembolization (DEB-TACE) compared with Conventional Transarterial Chemoembolization (cTACE) in patients with hepatocellular carcinoma (HCC) that is beyond the Milan criteria and who have previously undergone a Transjugular Intrahepatic Portosystemic Shunt (TIPS) procedure. The TIPS procedure is commonly performed to manage complications of portal hypertension, such as variceal bleeding or refractory ascites, in patients with cirrhosis. However, after TIPS, treatment options for HCC-particularly in cases exceeding the Milan criteria-remain limited and not well-defined in current guidelines.

While TACE is a standard locoregional therapy for intermediate-stage HCC, its application in patients with a prior TIPS is controversial due to altered hepatic hemodynamics, which may increase the risk of liver toxicity and compromise treatment safety and efficacy. Preliminary retrospective data suggest that DEB-TACE, which uses calibrated drug-eluting microspheres, may offer a safer and more effective alternative to cTACE in this specific patient population by providing more controlled drug delivery and potentially reducing systemic and hepatic toxicity.

The primary objective of this study is to determine whether DEB-TACE improves Overall Survival (OS) compared to cTACE in patients with beyond-Milan HCC after TIPS. Secondary objectives include comparing the safety profile, Progression-Free Survival (PFS), Objective Response Rate (ORR), Disease Control Rate (DCR), and Quality of Life (QoL) between the two treatment arms.

The study aims to enroll 206 participants who will be randomly assigned in a 1:1 ratio to receive either DEB-TACE or cTACE. The trial will include a 24-month recruitment period and a 24-month treatment and follow-up phase, with a total study duration of 48 months. By directly comparing these two TACE approaches in a prospectively defined and randomized setting, this study seeks to provide high-level evidence to guide the optimal locoregional treatment strategy for HCC patients with a history of TIPS placement.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or clinically confirmed primary hepatocellular carcinoma, beyond Milan criteria (single lesion >5 cm OR ≥3 lesions with at least one ≥3 cm). At least one intrahepatic measurable lesion with tumor burden ≤50%, no distant metastasis. No prior antitumor therapy within 12 months before enrollment.
2. underwent TIPS procedure for secondary prevention of variceal bleeding or refractory ascites. Confirmed patent TIPS at 1-month follow-up with portosystemic blood flow visible throughout the shunt and Doppler velocity > 60 cm/s.
3. child-Pugh class A or B.
4. estimated survival ≥3 months.
5. adequate organ function:Neutrophils ≥1.5 × 10⁹/L; Platelets ≥50 × 10⁹/L; Hemoglobin ≥90 g/L; Serum albumin ≥30 g/L; Bilirubin ≤50 μmol/L; AST/ALT ≤5 × upper limit of normal (ULN), ALP ≤4 × ULN; INR ≤2.3; Creatinine ≤1.5 × ULN.

Exclusion Criteria:

1. diffuse hepatic infiltration, unassessable lesions on imaging, or tumor burden >50%.
2. simultaneous portal vein branch tumor thrombus or main portal vein tumor thrombus.
3. underwent liver transplantation or antitumor therapy after TIPS placement.
4. contraindications to TACE (e.g., portosystemic shunt, hepatofugal blood flow, significant atherosclerosis).
5. presence of brain metastases.
6. Allergy to contrast agents.
7. pregnancy, breastfeeding, or planning pregnancy within 2 years.
8. co-infection with HIV or syphilis.
9. concurrent other malignancy or history of other malignancy within the past 5 years.
10. severe cardiac, renal, or other organ dysfunction.
11. active clinically severe infection > Grade 2 (per NCI-CTC v5.0).
12. psychiatric/psychological conditions that may impair informed consent.
13. participation in other drug clinical trials within 12 months prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 24 months
  Time interval from date of randomization until the date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time interval from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Tumor response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Defined as the proportion of patients achieving complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) according to mRECIST criteria.
Adverse event | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Defined as the occurrence of ≥ Grade 3 hematological or non-hematological toxicities, graded per CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiiated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China